CLINICAL TRIAL: NCT06565663
Title: Decision Making in Metoidioplasty and Phalloplasty Gender Affirming Surgery (MaPGAS)
Brief Title: MaPGAS Decision Making
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: University of Utah (Other); Dartmouth College (Other); National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Rachel A. Moses, Assistant Professor, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY02002174; 1R01DK137994-01 (NIH)
Record Dates: First submitted 2024-06-19; First posted 2024-08-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-11

CONDITIONS: Gender Dysphoria; Gender Dysphoria, Adult; Gender Incongruence; Transgenderism; Transsexualism; Transgender Persons; Phalloplasty
Keywords: Gender-Affirming Surgery; Sex Reassignment Surgery; Gender Reassignment Surgery; Phalloplasty; Metoidioplasty; Transmasculine; FTM; Gender Dysphoria; Transgender; Penile Reconstruction; Female-to-Male; Neophallus; Transsexual; Genital Reconstruction; Reconstructive Urology
MeSH Terms: conditions — Gender Dysphoria; Transsexualism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MaPGAS Decision Aid Intervention (Experimental): Participants in this arm will be provided with access to a novel, web-based decision aid designed for individuals considering MaPGAS. The decision aid includes interactive components, educational materials regarding surgical options, risks, benefits, and patient testimonials. Participants will have unlimited access to the decision aid for four weeks prior to their surgical consultation.
  Interventions: Behavioral: MaPGAS Decision Aid
- MaPGAS Usual Care (No Intervention): Participants in this arm will receive the standard pre-consultation care provided by their healthcare provider, which does not include access to the novel decision aid. Standard care may include informational brochures. This group serves to compare the outcomes of traditional decision-making processes with those who use the decision aid.

INTERVENTIONS:
Behavioral: MaPGAS Decision Aid — This intervention involves a novel, web-based decision aid tool specifically designed to support transgender and non-binary individuals assigned female at birth in making informed decisions about Metoidioplasty and Phalloplasty Gender Affirming Surgeries (MaPGAS). The tool includes comprehensive information on surgical options, risks, benefits, and medical illustrations to aid in aligning surgical decisions with the individual's personal values and goals.
  Other Names: Metoidioplasty and Phalloplasty Gender Affirming Surgery Web-Based Pictorial Decision Aid
  Arms: MaPGAS Decision Aid Intervention

SUMMARY:
The goal of this clinical trial is to test a new online tool designed to provide clear and understandable information to help individuals considering Metoidioplasty and Phalloplasty Gender Affirming Surgery (MaPGAS)make informed decisions

The main questions it aims to answer are:

* How user-friendly is the decision aid for individuals considering metoidioplasty and phalloplasty?
* Does using the decision aid reduce uncertainty and improve readiness for making surgery decisions compared to usual care?

Participants in this study will:

* Be randomly assigned to either 1) receive usual care or 2) test the web-based decision aid.
* Share their feedback on the tool's usability and its helpfulness in supporting decision-making.
* Complete surveys before and after using the decision aid to measure any changes in their decision-making process.

Researchers will compare participants who used the decision aid with those who received standard care to see if the decision aid reduces decisional uncertainty and improves readiness for surgery.

DETAILED DESCRIPTION:
This study aims to evaluate the usability, acceptability, and preliminary efficacy of a novel, web-based decision aid (DA) for Metoidioplasty and Phalloplasty Gender Affirming Surgeries (MaPGAS).

MaPGAS are increasingly performed to improve gender congruence and quality of life, however, patients face complex decisions which may impact fertility, urinary and sexual function. Existing decisional uncertainty among transgender and non-binary individuals considering MaPGAS highlights the need for effective decision support tools. Prior research indicates a gap in validated decision support, partly due to insufficient understanding of patient needs and a lack of published outcomes or guidelines. This study builds on preliminary work that identified key decision-making factors among patients and healthcare providers, leading to the development of a co-developed web-based MaPGAS picture DA prototype.

Cognitive interviews with both participants considering or post MaPGAS and healthcare providers will refine the decision tool. The study will also investigate the DA's implementation within clinical settings to understand optimal administration timing and its impact on shared decision-making processes.

This study will employ a mixed-methods approach and a prospective randomized controlled trial to assess the DA's usability and acceptability using the System Usability Scale and focus group feedback. Additionally, it aims to evaluate the DA's preliminary efficacy in reducing decisional conflict and improving decision readiness and shared decision-making quality compared to usual care. This will be measured using validated tools such as the Decisional Conflict Scale, Preparation for Decision Making Scale, and CollaboRATE measure, alongside semi-structured patient and provider interviews.

This research aims to addressing the decisional needs of transgender and non-binary individuals considering MaPGAS, aiming to empower them with the tools needed for making informed, value-congruent decisions regarding their surgical options.

ELIGIBILITY:
Inclusion Criteria:

* Assigned female on the original birth certificate.
* Self-identifies as transgender male and/or gender non-binary.
* Able to speak, read, and understand English at a sixth-grade level.
* Aged 18 or older.
* Resides in the USA.
* For decision aid refinement: Considering metoidioplasty or phalloplasty, or is post-operative.
* For intervention and control arm: Has a consultation scheduled for metoidioplasty or phalloplasty.

Exclusion Criteria:

* Participants involved in the initial tool refinement focus groups cannot participate in the intervention or control group to avoid contamination of the study outcomes.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender male and/or gender non-binary.
Enrollment: 140 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Decisional Conflict Scale (DCS) Score Change | Baseline (within 1-2 weeks prior to using the decision aid) and follow-up (immediately after decision aid use, approximately 2-4 weeks later).
  The Decisional Conflict Scale (DCS) is used to measure personal perceptions of uncertainty in choosing options, factors contributing to uncertainty such as feeling uninformed, unclear about personal values, and unsupported in decision making, and perceived effectiveness of decision making. A change in DCS scores from baseline (pre-decision aid exposure) to post-decision aid exposure will be assessed to determine the impact of the decision aid on reducing decisional conflict. Scores range from 0 [no decisional conflict] to 100 [extremely high decisional conflict].
Preparation for Decision Making (PrepDM) Scale Score Change | Baseline (within 1-2 weeks prior to using the decision aid) and follow-up (immediately after decision aid use, approximately 2-4 weeks later).
  The Preparation for Decision Making (PrepDM) scale assesses a patient's perception of how useful a health-related decision aid is in preparing them to make a health decision. It evaluates the perceived helpfulness of the decision aid in understanding treatment options, clarifying personal values for the decision, and feeling prepared to talk with their health provider about the decision. The change in PrepDM scores before and after decision aid exposure indicates the aid's efficacy in improving decision readiness. Higher scores indicate higher perceived level of preparation for decision making.

SECONDARY OUTCOMES:
CollaboRATE Score Change Post-Surgical Consultation | Within one week following the surgical consultation.
  The CollaboRATE score is a brief patient-reported measure assessing the extent of shared decision-making experienced during medical encounters. It focuses on three core aspects: the explanation of health issues, the elicitation of patient preferences, and the integration of these preferences into the decision-making process. A comparison of CollaboRATE scores between control and intervention groups after the surgical consultation will indicate the decision aid's impact on enhancing shared decision making. Higher scores represent more shared decision making; scores can range from 0-100.
System Usability Scale (SUS) Score | Immediately after using the decision aid (approximately 2-4 weeks from baseline)
  The System Usability Scale (SUS) Score is a reliable tool for measuring the usability of the web-based decision aid. It consists of a 10-item questionnaire with five response options for respondents ranging from 'Strongly agree' to 'Strongly disagree'. It is widely used in the domain of user experience and measures the overall perceived usability of the decision aid. Higher scores represent a higher perceived system usability; scores can range from 0-100.

OTHER OUTCOMES:
Qualitative Feedback from Cognitive Interviews | Post-decision aid use, and post-surgical consultation (dates vary, approximately 2-6 weeks from baseline).
  Qualitative feedback will be obtained through cognitive interviews with participants to refine the decision tool. This feedback will include participants' experiences using the tool, its clarity, relevance, and any suggestions for improvement. The interviews aim to capture in-depth insights into the decision aid's effectiveness and areas for enhancement.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel A. Moses, MD, MPH, Principal Investigator — Dartmouth-Hitchcock Clinic
Locations (2):
- United States (2):
  - Dartmouth College, Hanover, New Hampshire
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
The study plans to share de-identified individual participant data (IPD) that underlie the results reported in publications, as well as the data dictionaries defining each field in the set. Sharing these datasets will enable secondary analyses by other researchers, promoting transparency and accelerating knowledge discovery in the field of gender affirming surgeries. The shared IPD will include demographic information, responses to surveys, and outcome measures such as the Decisional Conflict Scale, Preparation for Decision Making Scale, CollaboRATE measure, and other relevant data collected throughout the study.
Time Frame: The shared IPD and supporting documentation will become available starting 6 months after the publication of the main findings from the final dataset or two years from study completion, whichever comes first. The availability period for accessing these data will extend for five years, ensuring ample time for interested researchers to conduct secondary analyses.
Access Criteria: Access to the shared IPD will be granted upon request to researchers who provide a methodologically sound proposal intended for non-commercial purposes. Requests will be reviewed by the study team. Criteria for reviewing requests will include the scientific rationale, methodological approach, and the potential contribution to understanding or improving gender affirming surgeries. Approved researchers will be required to sign a data access agreement to ensure the confidentiality and proper use of the data.
  Information about how to request access to the IPD, including details of the review process and access criteria, will be made available on the study's dedicated webpage hosted by Dartmouth-Hitchcock Clinic's institutional repository, Dataverse.